CLINICAL TRIAL: NCT06179654
Title: Preoperative Pelvic Floor Physical Therapy to Minimize Stress Urinary Incontinence After Holmium Laser Enucleation of the Prostate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Smita De, Staff Urologist, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-1128
Record Dates: First submitted 2023-11-29; First posted 2023-12-22 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Benign Prostatic Hyperplasia With Outflow Obstruction; Urinary Retention; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Urinary Retention; Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: 2-cohort study. Group A will start pelvic floor exercises before surgery and Group B will start exercises after surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preoperative PFPT (Experimental): This group of patients will be instructed to start pelvic floor physical therapy 1 month before surgery.
  Interventions: Behavioral: Preoperative pelvic floor physical therapy
- Postoperative PFPT (No Intervention): This group of patients will be instructed to start pelvic floor physical therapy after surgery (standard of care).

INTERVENTIONS:
Behavioral: Preoperative pelvic floor physical therapy — Pelvic floor physical therapy to start before prostate surgery rather than after surgery.
  Arms: Preoperative PFPT

SUMMARY:
The purpose of this study is to allow us to assess the effectiveness (or success) of starting pelvic floor physical therapy (i.e. exercises for your pelvic muscles) prior to HoLEP (holmium laser enucleation of the prostate) surgery for enlarged prostates in order to manage or prevent urinary incontinence (i.e. leaking) after surgery (i.e. post-operatively). Your pelvic floor refers to the muscles under your bladder along your pelvic bones that prevent you from leaking urine or stool. Traditionally, pelvic floor physical therapy is started after surgery and continued until urinary continence (i.e. no leaking of urine) is regained. We want to assess if beginning pelvic floor physical therapy prior to surgery (and continuing afterwards) reduces the time required to regain urinary continence following HoLEP.

DETAILED DESCRIPTION:
The incidence of benign prostatic hyperplasia (BPH) in men significantly increases with age and is estimated to impact over 80% of men 70 to 80 years of age. HoLEP is one of many treatments for BPH and associated lower urinary tract symptoms. Compared to other minimally invasive surgical techniques for treatment of BPH, HoLEP has been found to have superior outcomes and is a prostate size-independent procedure with excellent durability, high efficacy, and low complications rates. However, transient stress urinary incontinence (SUI) following HoLEP may last for several months after surgery and can lead to diminished patient quality of life during the recovery period. Measures to prevent or reduce post-operative SUI following HoLEP, including PFPT, may improve patient outcomes.

SUI is also commonly documented after radical prostatectomy (RP) for prostate cancer. The mechanism for incontinence in both RP and HoLEP is thought to at least partially be related to temporary weakness of the external urinary sphincter, which is part of the pelvic floor musculature. While it is unclear if post-operative PFPT alone reduces SUI for patients who have undergone RP, there is evidence that PFPT started pre-operatively and continued post-operatively can decrease SUI following RP.

The utilization of pre-operative PFPT for patients undergoing HoLEP to reduce post-operative SUI is currently not well documented. To date, only one study has demonstrated evidence that PFPT prior to HoLEP may improve continence at 3 months. However, the study included patients with a BMI significantly lower than average in the United States, utilized an unclear PFPT program, and had a relatively small median prostate size (~60 mL), which is important as studies have shown that prostate size can affect post-operative incontinence.

We propose a prospective randomized trial to investigate the efficacy of standardized pre-operative PFPT in reducing SUI and improving patient QoL following HoLEP. This study will help determine the role of pre-operative PFPT in the management of HoLEP associated SUI.

ELIGIBILITY:
Inclusion Criteria:

1. Age: >=18 years of age
2. Sex: male sex assigned at birth (needs to have a prostate)
3. BMI: all BMI
4. Ethnic background: all ethnicities
5. Medical history: patients scheduled to undergo HoLEP for BPH/LUTS and associated complications (i.e. gross hematuria, retention, etc.).

Exclusion Criteria:

1. Neurological disorders: patients with a history of a neurologic disorder that could affect muscle function, neurogenic bladder, lumbosacral spine pathology
2. Specific urologic conditions: patients with pre-operative indwelling catheter, urethral stricture greater than 1 centimeter in length or requiring dilation/incision, indwelling ureteral stent
3. History of pelvic radiation: patient with prior pelvic radiation will be excluded
4. Patients unable to give consent
5. Non-English speaking patients given the need for multiple surveys and telephone follow-ups.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Time to continence | 6 months after surgery
  Time to recover from transient postoperative stress urinary incontinence

SECONDARY OUTCOMES:
Uroflow | 6 months after surgery
  urine flow rate (milliliters/second)
Post void residual | 6 months after surgery
  Residual urine after voiding (milliliters)
international prostate symptom score | 6 months after surgery
  validated questionnaire on urination symptoms
operative time | day of surgery
  length of surgery (minutes)
length of stay | 30 days after surgery
  days of hospitalization after surgery
catheter duration | 30 days after surgery
  days with catheter after surgery
infectious complications | 30 days after surgery
  urinary tract infection complication after surgery
emergency room visits | 30 days after surgery
  number of emergency room visits related to surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No